CLINICAL TRIAL: NCT05567484
Title: Comparative Study Between Pulsed and Continuous Itraconazole for the Treatment of Onychomychosis
Brief Title: Comparative Study Between Pulsed and Continuous Itraconazole for the Treatment of Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Rohida Rahmat, principle investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMH Abbottabad
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Onychomychosis
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A pulse thearpy of itraconazole (Active Comparator): Patients in pulse therapy group received oral itraconazole 100 mg, two capsules twice daily for seven days a month
  Interventions: Drug: Itraconazole
- Group B continous thearpy of itraconazole (Active Comparator): Patients in continuous therapy group, received continuous oral 100 mg of itraconazole once daily for 12 weeks continuously.
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — 100 mg two capsules of itraconazole were given twice daily to 30 patient group A for one week per month.baseline LFTs were also monitered
  Other Names: capsule icon

SUMMARY:
The term onychomycosis is used for a chronic fungal infection of the nail which when caused by dermatophytes, becomes tinea unguium. It not only includes the dermatophytes but also saprophytic molds infections and yeasts. Thorough literature research has revealed that 90% toenail and 75% fingernail onychomycosis are a result of dermatophytes arguably by Trichophyton mentagrophytes and Trichophyton rubrum. Comorbid conditions such as diabetes mellitus and peripheral arterial disease and immunosuppression due to HIV plays a catalytic role in its prognosis. In a study, upon comparison of placebo with continuous terbinafine 250 mg daily for 24 weeks and continuous terbinafine 250 mg daily for 16 weeks, no significant differences were observed by the researchers between the two methods i.e continuous and pulse regimens of terbinafine, itraconazole, and fluconazole respectively. Moreover, in one another research study, the researchers also did not find significant superiority of continuous itraconazole 200 mg daily for 12 weeks over pulsed itraconazole 400 mg in the treatment of terms onychomycosis of mycological cure that is the reason why continuous daily itraconazole 200 mg for 24 weeks has so far performed best in rank probabilities over other therapies, but its clinical significance is still debated. The purpose of carrying out this study was to carry out comparison between pulsed and continuous itraconazole for the treatment of onychomycosis as previous literature shows ambiguous results, therefore, this study will cement the rare evidence pertaining to the efficacy of pulsed and continuous itraconazole in the treatment of onychomycosis in our local population

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20-60 years
* Patients positive for fungus via direct microscopy due to the identification of hyphae or blastospores on the target toenail
* Patients positive fungal culture. Patients who had not applied any topical agent to the target toenail for the last 1 month

Exclusion Criteria:

* Pregnant patients
* Patients with poor adherence
* Lactating women.
* Patients previously allergic to oral itraconazole.
* Patients with elevated baseline liver function tests such as ALT, AST, alkaline phosphatase, and total bilirubin twice the upper limit of normal
* History of renal disease.
* Patients unresponsive to systemic antifungal therapy within the past year
* History of using systemic immunosuppressants.
* Patients exhibiting evidence of ventricular dysfunction and history of congestive heart disease
* Immunocompromised patients

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
effectiveness of pulse therapy of itraconazole and continuous therapy of itraconazole for the treatment of onychomycosis as assessed by ONYCHOMYCHOSIS SEVERITY INDEX (OSI) | 12 weeks
  Onychomycosis severity index was used to measure the effectiveness of drug

CONTACTS AND LOCATIONS:
Locations (1):
- cmh Abbottabad, Abbottabad, Khyber Pakhtunkhwa, Pakistan